CLINICAL TRIAL: NCT01295658
Title: Cancer Survivor Registry: The Breast Cancer M.A.P. (Mind Affects the Physical) Project
Status: Completed | Type: Observational
Sponsor: Cancer Support Community, Research and Training Institute, Philadelphia (Other)
Responsible Party: Principal Investigator, Elissa Kranzler, PhD, Director of Research, Cancer Support Community, Cancer Support Community, Research and Training Institute, Philadelphia
Other Study IDs: CSC-MAP-0102
Record Dates: First submitted 2011-02-11; First posted 2011-02-14 (Estimated); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Cancers
Keywords: cancer; cancer survivorship; psychosocial needs; cancer experience; metastatic breast cancer; breast cancer; caregiver
MeSH Terms: conditions — Neoplasms; Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cancer Survivors: This is a broad observational study conducted online at www.cancerexperienceregistry.org, or via pen and paper survey obtained by calling the cancer support helpline at 888-793-9355
  Any individual who has ever received a cancer diagnosis, regardless of disease type, stage, treatment, and time since diagnosis, can take part in this study.

SUMMARY:
Cancer Survivor Registry: The Breast Cancer M.A. P. (Mind Affects the Physical M.A.P.) Project to identify and help us understand the emotional and social needs of breast cancer survivors.

DETAILED DESCRIPTION:
The Cancer Survivor Registry: The Breast Cancer M.A.P. (Mind Affects the Physical) Project was the first registry of its kind to look at the emotional and social needs of individuals diagnosed with breast cancer and track how their needs changed throughout their cancer journey. Data will raise awareness and help develop programs to address the needs of breast cancer survivors. Findings from the Registry are disseminated online at www.CancerSupportCommunity.org/RegistryIndexReport2017

ELIGIBILITY:
Inclusion Criteria:

* Having received a cancer diagnosis

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Any individual who has received a cancer diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 3729 (Actual)
Dates: Start 2010-05 (Actual); Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Self-reported quality of life measures | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Linda House, RN, BSN, MSM, Principal Investigator — Cancer Support Community
Locations (1):
- Cancer Support Community Research & Training Institute, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Cancer Experience Registry: An Online Initiative to Change the Future of Cancer Care — http://www.cancerexperienceregistry.org